CLINICAL TRIAL: NCT00118222
Title: A Randomized Prospective Two Arm Clinical Trial of High Light Dose And Low Light Dose PDT in the Treatment of Recurrent Malignant Supratentorial Gliomas Using Porfimer Sodium [Photofrin]
Brief Title: High Light and Low Light Dose PDT in Glioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert Maciunas, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU4303; P30CA043703 (NIH); CASE-4303 (Other: Case Comprehensive Cancer Center); CWRU-00003937; CWRU-4303 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult mixed glioma; adult anaplastic astrocytoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioma; Astrocytoma; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Dihematoporphyrin Ether; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low light dose during surgery (Active Comparator): Arm I: During surgery, patients receive low light dose photodynamic therapy.
  Interventions: Drug: porfimer sodium; Procedure: adjuvant therapy; Procedure: conventional surgery
- High light dose during surgery (Active Comparator): Arm II: During surgery, patients receive high light dose photodynamic therapy.
  Interventions: Drug: porfimer sodium; Procedure: adjuvant therapy; Procedure: conventional surgery

INTERVENTIONS:
Drug: porfimer sodium — All patients receive porfimer sodium IV.
  Other Names: dihematoporphyrin ether; Photofrin II; Porfimer
Procedure: adjuvant therapy — All patients receive porfimer sodium IV.
  Other Names: dihematoporphyrin ether; Photofrin II; Porfimer
Procedure: conventional surgery — All patients receive porfimer sodium IV. One day later, patients undergo craniotomy and tumor resection.

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as porfimer sodium, that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. Giving photodynamic therapy after surgery may kill any remaining tumor cells.

PURPOSE: This randomized clinical trial is studying two different light doses of photodynamic therapy using porfimer sodium to compare how well they work in treating patients who are undergoing surgery for recurrent malignant astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival of patients undergoing surgical resection for recurrent high-grade malignant supratentorial astrocytoma treated with intraoperative high vs low light dose photodynamic therapy using porfimer sodium.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

All patients receive porfimer sodium IV. One day later, patients undergo craniotomy and tumor resection.

* Arm I: During surgery, patients receive low light dose photodynamic therapy.
* Arm II: During surgery, patients receive high light dose photodynamic therapy. After completion of study treatment, patients are followed at 1 day, 6 weeks, and 3 months and then every 3 months for up to 2 years.

PROJECTED ACCRUAL: Approximately 120 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant supratentorial astrocytoma, glioblastoma, or mixed oligo-astrocytoma

  * Grade 3 or 4 tumor, defined as presence of ≥ 2 of the following features:

    * Nuclear atypia
    * Mitosis
    * Endothelial proliferation
    * Necrosis
* Recurrent disease

  * Failed prior surgery and radiotherapy
* Tumor suitable for radical resection by imaging studies

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing to avoid direct sun-light exposure for 6 weeks after photodynamic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Time to progression and survival measured | at 4-6 weeks post-operatively and then every 3-4 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Maciunas, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States